CLINICAL TRIAL: NCT02010541
Title: The Influence of Diabetes Related Technology, Education and Psychological Support on Metabolic Control in Young Children With Type 1 Diabetes
Brief Title: The Influence of Technology, Education and Psychological Support on Metabolic Control in Children With T1D
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: Slovenian Research Agency (ARRS) (Unknown)
Responsible Party: Principal Investigator, Tadej Battelino, Head, Dept. of Pediatric Endocrinology, Diabetes & Metabolism, University Children's Hospital, UMCL, University Medical Centre Ljubljana
Other Study IDs: TECH-EDU-KIDS-T1D-2013
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes among young children, sensor, insulin pump, education, psychological support
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- insulin pump group: 20 children below the age of 7 years who use an insulin pump for at least 6 months, more than 6 months of duration of type 1 diabetes, complete remission, no associated disease (normal blood pressure for age, only therapy insulin).
- RT (real time) -CGMS group: 20 children below the age of 7 years who use an insulin pump and RT-CGMS on regular basis for at least 6 months, more than 6 months of duration of type 1 diabetes, complete remission, no associated disease (normal blood pressure for age, only therapy insulin). pump for at least 6 months, and children below the age of 7 years who use RT-CGMS on regular

SUMMARY:
The first purpose of this study is to is to compare metabolic control of type 1 diabetes among children under the age of 7 years who use an insulin pump and a real-time (RT) glucose sensor, and children who use only insulin pump; the investigators will also determine dietary habits, their knowledge of type 1 diabetes management and emotional aspects of experiencing illness in the family, in both groups of children.

ELIGIBILITY:
Inclusion Criteria:

* age up to 7 years
* insulin pump for at least 6 months
* more than 6 months of duration of type 1 diabetes
* complete remission
* normal blood pressure for age, only therapy insulin.

Exclusion Criteria:

* age over 8 years
* type 1 diabetes less than 6 months
* insulin pump less than 6 months
* still in remission
* associated diseases on drug therapy, high blood pressure

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children that have diabetes in Slovenia are controlled at the Dept. of Pediatric Endocrinology, Diabetes & Metabolism, University Children's Hospital, UMCL and the population will be taken from here
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-04 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Glycaemic control | 3 months
  We will determine HbA1c, average blood glucose, number of blood glucose readings/use of sensors, average AUC for sensor users, readings above and under target for both groups at the beginning and afer 3 months.

SECONDARY OUTCOMES:
knowledge on diet and diabetes management | 3 months
  Questionnaire on diet, questionnaire on diabetes management; we will assess the knowledge on diet in T1D and diabetes management in both groups at the beginning, we will give support wherever needed and check after 3 months if it had an influence on metabolic control.

OTHER OUTCOMES:
Number of adverse events | 3 months
Quality of Life measures | 3 months
  CBCL 1 ½-5 or CBCL 6-18 questionnaire, PSI questionnaire, Experiences in Close Relationships- Relationship Structures questionnaire; we will assess if the psychological issue is an important factor in diabetes management

CONTACTS AND LOCATIONS:
Overall Officials: Tadej Battelino, Study Chair — Dept. of Pediatric Endocrinology, Diabetes & Metabolism, University Children's Hospital, UMCL
Locations (1):
- Dept. of Pediatric Endocrinology, Diabetes & Metabolism, University Children's Hospital, UMCL, Ljubljana, Slovenia